CLINICAL TRIAL: NCT02992444
Title: Evaluation of the Influence of Output on Skin Covered by Adhesives (Round 5)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_05
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2017-01

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 5 (Experimental): This is a sub-study testing the effect of real output applied under two adhesive strips on the skin after 8 hours.
  There is one visit:
  Two adhesive strips (standard adhesive strip and Experimental adhesive strip)are applied on the peristomal skin and allowed to sit for 8hours before being removed.
  Interventions: Other: Standard adhesive strip; Other: Experimental adhesive strip

INTERVENTIONS:
Other: Standard adhesive strip — This is a standard adhesive strip (hydrocolloid)
Other: Experimental adhesive strip — This is a strip of a newly developed adhesive.

SUMMARY:
This study investigates the impact real output has on peristomal skin covered by an adhesive

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had an ileostomy for more than one year
4. Have intact skin on the area used in the evaluation
5. Has an ileostomy with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Participating in other interventional clinical investigations or have previously participated in this evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 4 - 24 hours
  The skins barrier function is measured using trans epidermal water loss after removing the adhesive from the skin

CONTACTS AND LOCATIONS:
Overall Officials: Lene Feldskov, M. Sci, Principal Investigator — Senior R&D Scientist
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No